CLINICAL TRIAL: NCT06701890
Title: Observational Study of Travellers Pathologies
Acronym: EOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-069; 2023-A02574-41 (Other: ID-RCB number)
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Travel-Related Illness
Keywords: Travel; Risk Factors; Pathology; Arbovirose
MeSH Terms: conditions — Travel-Related Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults planning to travel outside metropolitan France. (Experimental): Human biological samples :
  * Blood sample
  * fecal sample
  Interventions: Other: Blood sample collection; Other: Fecal sample collection

INTERVENTIONS:
Other: Blood sample collection — 16 mL at inclusion 16 mL at 1 month after return from travel
Other: Fecal sample collection — 1 sample at inclusion
  1 sample at day 1, day 7, day 14, day 21, 1 month and 2 month after return from travel

SUMMARY:
Traveling to emerging countries is associated with a significant risk of encountering health issues specific to the destination, such as gastrointestinal and respiratory infections, malaria episodes, and road traffic accidents.These conditions are associated with behavioral, geographical, or environmental risk factors. A better understanding of these factors will enable the development of targeted recommendations to minimize travel related health issues.

The main objective of this study is to determine the incidence of pathologies occurring during travel outside the metropolitan territory.

DETAILED DESCRIPTION:
Traveling to emerging countries is associated with a significant risk of encountering health issues specific to the destination, such as gastrointestinal and respiratory infections, malaria episodes, and road traffic accidents.These conditions are associated with behavioral, geographical, or environmental risk factors. A better understanding of these factors will enable the development of targeted recommendations to minimize travel related health issues.

The main objective of this study is to determine the incidence of pathologies occurring during travel outside the metropolitan territory.

Furthermore, two key aspects from a Public Health perspective are associated with travel and the globalization of exchanges: the acquisition of emerging pathogens or pathogens with antimicrobial resistance of concern.

To study these two aspects, the EOP study includes two sub-studies called EOP-Arbo and EOP-AMR.

* EOP-Arbo : The objective of this sub-study is to determine the risk of contracting an arboviral disease during travel, as well as the factors that may favor infection. For this, blood samples will be collected.
* EOP-AMR : The objective of this sub-study is to determine the risk of contracting an antibiotic-resistant bacteria during the trip. For this, faecal samples will be collected.

ELIGIBILITY:
1. Inclusion Criteria :

   1. For all participants in the EOP study :

      * Major subject (age ≥ 18)
      * Owns a smartphone compatible with electronic data collection
      * Preparing to travel outside mainland France
      * Affiliated with or covered by Social Security or private insurance
      * Willing to participate in the EOP study
   2. For the EOP-Arbo Sub-study :

      - Subject who has consented to participate in the EOP_Arbo study.
   3. For the EOP-AMR Sub-study :

      * Subject who has consented to participate in the EOP_AMR study.
2. Exclusion Criteria:

   1. For all participants in the EOP study :

      * Travel duration ≤ 3 days
      * Travel duration > 12 months
      * Person traveling as part of an expatriation without planned movement outside the settlement in the destination country
      * Person under legal protection or unable to express consent for participation
   2. For the EOP-Arbo Sub-study :

      - Individuals deemed clinically and/or biologically unfit by the investigator to undergo the blood samples required for the study.
   3. For the EOP-AMR Sub-study :

      * No specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11000 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2034-12 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
Determine the incidence of pathologies occurring during a travel outside the metropolitan territory. | 10 years
  Number of subjects who developed a pathology during the travel among participants

SECONDARY OUTCOMES:
For EOP-Arbo sub-study : Determine the prevalence for the occurrence of an arboviral disease (dengue, chikungunya, Zika) during the travel. | 10 years
  Number of arboviral diseases (dengue, chikungunya, Zika) during the travel among participants
For EOP-AMR sub-study : Determine the prevalence for the acquisition of multi-resistant bacteria (MRB) during the travel. | 10 years
  Proportion of subjects with multi-resistant bacteria acquired during the travel

CONTACTS AND LOCATIONS:
Overall Officials: Fabien TAIEB, MD, Principal Investigator — Medical Center of Institut Pasteur
Locations (1):
- Medical Center of Institut Pasteur, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided